CLINICAL TRIAL: NCT05595434
Title: Study of Reality-monitoring Process and Influence of Stress Using an Electrophysiological Approach
Brief Title: Reality-monitoring & Stress
Acronym: REALIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-A01390-43
Record Dates: First submitted 2022-10-13; First posted 2022-10-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: reality-monitoring; stress

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind study including 40 healthy subjects who will be randomly divided into 2 groups.
Who Masked: Participant
Masking Description: Participants will not be informed about the nature (active or placebo) of the stress test they will perform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stress group (Experimental): 20 healthy subjects will be subject to the active condition of a standardized stress protocol
  Interventions: Procedure: Acute Maastricht Stress Test (MAST), active condition.
- placebo stress group (Placebo Comparator): 20 healthy subjects will be subject to the placebo condition of a standardized stress protocol.
  Interventions: Procedure: Acute Maastricht Stress Test (MAST), placebo condition

INTERVENTIONS:
Procedure: Acute Maastricht Stress Test (MAST), active condition. — The MAST is a standardized stress protocol combining a 5 min preparation phase and 10 min acute stress phase. The last phase is composed by an alternation of physical and psychosocial stressors. In the active condition, participants have to switch between immersion of the hand into cold water and complex mental arithmetic operations.
  Arms: active stress group
Procedure: Acute Maastricht Stress Test (MAST), placebo condition — The MAST is a standardized stress protocol combining a 5 min preparation phase and 10 min acute stress phase. The last phase is composed by an alternation of physical and psychosocial stressors. In the placebo condition, participants have to switch between immersion of the hand into tempered water and simple mental arithmetic counts.
  Arms: placebo stress group

SUMMARY:
Reality-monitoring is a crucial cognitive process in daily life to remember the source of an information. Deficits of reality-monitoring have been shown into the continuum of schizophrenia, suggesting a preexisting alteration in population at-risk for psychosis that will be exacerbated during psychotic transition. It is admitted that stress plays a crucial role in the psychotic transition and can alter cognitive performances. However, less is known about the effects of stress on reality-monitoring, even though this process appears to be central in psychotic disorders.

The aim of this project is to investigate the effect of stress on reality-monitoring, both on behavioral and neurophysiological aspects

DETAILED DESCRIPTION:
Forty healthy subjects will be included in the study. Participants will be subject to a standardized stress protocol, half of them receiving an active stress and the other half receiving a placebo. All participants will also complete a reality-monitoring task, electrophysiological (EEG) recordings as well as socio-demographic and psychometric evaluations

ELIGIBILITY:
Inclusion Criteria:

* Right-handed Men and Women aged between 18 and 30
* Having given their written informed consent
* For women: oral contraceptive use
* French speakers and readers

Exclusion Criteria:

* Do not consent to be included in the study
* Smokers
* Night workers
* Having visual or hearing impairments that could prevent the successful completion of tasks involving reading or listening to sounds
* Taking drug treatment (except oral contraceptive)
* Having a somatic pathology in particular neurological, endocrinal or blood circulation diseases (e.g., Raynaud's disease)
* Having personal or first-degree relatives' history of diagnosed psychiatric disorders (according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - DSM5)
* Having psychotic prodomes measured by a score above 6 in the "prodomal questionnaire' - PQ-16 (Ising et al., 2012)
* Having developed musical abilities (that is, regularly practicing a musical instrument)
* Being pregnant or nursing

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Reality-monitoring performances | within 1 hour after the stress procedure
  scores obtained at the reality-monitoring task (accuracy, range 0-100%)

SECONDARY OUTCOMES:
electroencephalogram (EEG) activity | 1time within 1 hour after the stress procedure
  EEG activity recorded at rest (spectral power) and during reality-monitoring task
Working memory | 1 time within 1 hour after the stress procedure
  scores at the n-back task (expressed as % of good responses)
Basic auditory performances | 1 time within 1 hour after the stress procedure
  scores at the Tone Matching Task (expressed as % of good responses)
Salivary cortisol | throughout and within 1 hour after the stress procedure
  Salivary cortisol (in µg/L)
Blood pressure | throughout and within 1 hour after the stress procedure
  blood pressure (both systolic and diastolic, in mmHg)
Heart rate | throughout and within 1 hour after the stress procedure
  Heart rate (in beats per minute)
expression rate of genes involved in the regulation of the glucocorticoid receptor signaling pathway | 1 time before and 1 time 1 hour after the stress procedure
  The expression rate of genes of the glucocorticoid receptor signaling pathway (NR3C1, FKBP4, HSP90, HSP70, FKBP5, BAG1, PTGES3)
Subjective stress | 1 time before and 1 time 1 hour after the stress procedure
  Subjective stress assessed with the STAI-YA (scores between 20 and 80)
Psychometric characteristics that may influence stress response (1) | Basline, before the stress procedure
  Scores at the 16-item Prodromal Questionnaire (PQ-16), ranging between 0 and 16 (higher scores indicate higher psychotic risks).
Psychometric characteristics that may influence stress response (2) | Basline, before the stress procedure
  Scores at the Childhood Trauma Questionnaire (CTQ), between 28 and 140 (higher scores indicate higher trauma exposure)
Psychometric characteristics that may influence stress response (3) | Basline, before the stress procedure
  State Trait Anxiety Inventory (form B) scores between 40 and 160 20 and 80 (STAI-YB) between 20 and 80 (higher scores indicate higher state anxiety)
Psychometric characteristics that may influence stress response (4) | Basline, before the stress procedure
  Scores at the Schizotypal Personality Questionnaire (SPQ), between 0 and 74 (higher scores indicate higher schizotypal traits)
Psychometric characteristics that may influence stress response (5) | Basline, before the stress procedure
  Scores at the Launay-Slade Hallucinations Scale (LSHS), between 0 and 64 (higher scores indicate a greater likelihood of experiencing hallucinations)

CONTACTS AND LOCATIONS:
Overall Officials: Mondino Marine, PhD, Principal Investigator — hospital le vinatier
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France